CLINICAL TRIAL: NCT01129752
Title: The Neural Correlates of Mood and Cognitive Bias in a Population at Risk for Depression: Maternal Cognitive and Emotional Functioning
Brief Title: Mothers With a History of Depression and Their 10-14 Year Old Daughters
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Ian H. Gotlib, Principal Investigator, Stanford University School of Medicine
Other Study IDs: SU-03172010-5264; 13058
Record Dates: First submitted 2010-05-21; First posted 2010-05-25 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Depression; Depressive Disorder, Major
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All participants are asked to submit saliva samples during their second session using sterile salivette containers in order to assess cortisol levels. There is no risk involved in giving these samples.

GROUPS / COHORTS (1):
- children at risk for depression: children at familial risk for depression
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — there is no intervention for this study

SUMMARY:
The purpose of this study is to investigate risk factors associated with depression and how such factors might be transmitted cross-generationally. The investigators are conducting an integrative assessment of emotion regulation and stress reactivity in a group of mothers with and without a history of depression and their daughters.

DETAILED DESCRIPTION:
The purpose of this study is to investigate risk factors associated with depression and how such factors might be transmitted cross-generationally. We are conducting an integrative assessment of emotion regulation and stress reactivity in a group of mothers with and without a history of depression and their daughters. We use a range of methodologies to evaluate these processes, including self-report measures, information-processing performance, HPA-axis functioning and reactivity, and neural responses to emotional stimuli following exposure to stressful experiences.

ELIGIBILITY:
Inclusion Criteria:

* Eligible mothers must read and speak English fluently and have a child between the ages of 9 and 15 years old.
* Mothers must either have no history of psychopathology or have a history of depression during their child's lifetime.

Exclusion Criteria:

* Eligible mothers cannot:

  * currently be in treatment for drug or alcohol abuse
  * have significant symptomatology related to psychopathology outside of depression
  * have a medical history of neurological injury or impairment.
* Mothers who meet the requirements for inclusion in the control group must not have a history of any Axis I disorder.

Ages: 9 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Eligible mothers must read and speak English fluently and have a child between the ages of 9 and 15 years old. Mothers must either have no history of psychopathology or have a history of depression during their child's lifetime.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2004-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Onset of depression | 18 months
  participants are interviewed in an 18-month follow-up session

CONTACTS AND LOCATIONS:
Overall Officials: Ian H Gotlib, PhD, Principal Investigator — Stanford University Department of Psychology
Locations (2):
- United States (2):
  - Stanford University Department of Psychology, Stanford, California
  - Stanford University School of Medicine, Stanford, California